CLINICAL TRIAL: NCT06864780
Title: Comparative Study on the Effectiveness of Posture Correction Exercises for Forward Head Posture in Chronic Smartphones and Laptop Users.
Brief Title: Posture Correction Exercises for Forward Head Posture in Chronic Smartphone and Laptop Users
Acronym: Comparative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/01008-Hafsa Rahim
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Forward Head Posture
Keywords: Forward Head Posture (FHP)
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Analgesia; Posture

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Masking Description: This study follows an analytical research model designed to compare the effectiveness of different posture correction exercises in treating Forward Head Posture (FHP) among frequent smartphone and laptop users. The model includes key components such as participant selection, intervention methods, data collection, and statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Posture Correction Exercises
  Usage of modalities like hot pack & TENS along with the following exercises:
  1. Chin Tucks (Seated or standing, retracting the chin while keeping eyes level)
  2. Cervical Retraction with Resistance Band (Pull band backward while maintaining retracted chin position)
  3. Shoulder Blade Squeeze (Seated or standing, squeeze shoulder blades together)
  4. Wall Posture Alignment (Standing against the wall, maintaining a neutral spine and retracting the head)
  Interventions: Other: Posture Correction Exercises; Other: Strengthening and Stretching Exercises
- Group B (Experimental): Strengthening and Stretching Exercises
  Usage of modalities like hot pack & TENS along with the following exercises:
  Upper Trapezius Stretch (Lateral neck stretch to release tightness) Levator Scapulae Stretch (Tilting head diagonally downward while applying gentle pressure) Deep Neck Flexor Strengthening (Supine, lifting head slightly while maintaining retraction) Scapular Retraction with Resistance Band (Seated or standing, pulling band while squeezing shoulder blades)
  Interventions: Other: Posture Correction Exercises; Other: Strengthening and Stretching Exercises

INTERVENTIONS:
Other: Posture Correction Exercises — This intervention focuses on improving forward head posture (FHP) through a series of corrective exercises aimed at enhancing cervical alignment, reducing muscle strain, and reinforcing proper posture habits. The exercises include chin tucks, cervical retraction with resistance bands, shoulder blade squeeze, and wall posture alignment. Participants will receive hot pack therapy (15-20 mins) for cervical muscle relaxation and TENS (10 mins) for pain relief before and after exercises. These exercises target deep cervical flexors and postural stabilizers to help retrain the neck and upper back muscles, promoting long-term postural correction. The intervention will be performed 3 times per week for 6 weeks under supervision, with a focus on maintaining correct postural alignment during daily activities.
  Other Names: Hot Pack (15-20 min) & TENS (10 min) for relaxation and pain relief, followed by corrective exercises to improve cervical alignment and posture
Other: Strengthening and Stretching Exercises — This intervention aims to address muscle imbalances associated with forward head posture (FHP) by incorporating stretching of tight muscles (upper trapezius, levator scapulae) and strengthening of weak postural muscles (deep neck flexors, scapular stabilizers). The exercises include upper trapezius stretch, levator scapulae stretch, deep neck flexor strengthening, and scapular retraction with resistance bands. Participants will undergo hot pack therapy (15-20 mins) for cervical muscle relaxation and TENS (10 mins) for pain relief before and after exercises. The stretching exercises will help release tension in overactive muscles, while strengthening exercises will restore muscular balance, improving posture and reducing neck discomfort. The intervention will be conducted 3 times per week for 6 weeks with supervised sessions to ensure proper technique and progressive improvement in flexibility and strength.
  Other Names: Hot Pack (15-20 min) & TENS (10 min) for relaxation and pain relief, followed by stretching tight muscles and strengthening weak postural muscles.

SUMMARY:
This study aims to compare different posture correction exercises to see which is most effective in improving forward head posture (FHP) in people who frequently use smartphones and laptops. FHP occurs when the head leans forward, putting extra strain on the neck and shoulders, leading to discomfort and pain. With the increasing use of digital devices, many individuals experience posture-related issues without realizing their long-term effects. This study will assess the impact of specific exercises, such as chin tucks and neck isometric holds, in realigning the head and relieving discomfort. The research will involve 56 participants aged 18-40 who use their devices for at least 2-3 hours daily. Participants will perform targeted exercises over four weeks, and improvements in posture and pain levels will be measured using a standardized scale. The study aims to determine whether structured posture correction exercises can help alleviate FHP and improve overall well-being in frequent digital device users.

DETAILED DESCRIPTION:
This study focuses on understanding and improving Forward Head Posture (FHP), a common problem seen in people who frequently use smartphones and laptops. FHP occurs when the head moves forward beyond its natural alignment, causing excessive strain on the neck, shoulders, and upper back. It can lead to pain, stiffness, headaches, and long-term postural problems. With the increasing use of digital devices, more people-especially young adults-are experiencing FHP without realizing its impact on their health. This study aims to compare different posture correction exercises to determine which is most effective in reducing FHP and associated discomfort. People often use smartphones and laptops for long hours without paying attention to their posture. Research shows that prolonged device use can cause poor posture habits, leading to musculoskeletal issues over time. If left untreated, FHP can contribute to chronic neck pain, reduced mobility, and even long-term spinal problems. This study is important because it will help identify simple exercise-based solutions that can improve posture and reduce discomfort. The findings can benefit smartphone and laptop users by promoting awareness and encouraging healthy posture habits.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Demographic criteria; age from 18-40 years both male & female.
* Smartphone usage for minimum of 2-3 hours daily from last one year
* Willingness to participate.
* No previous treatment for forward head posture.

Exclusion Criteria:

* Participants who fall in this category would be excluded of the study.
* Spinal deformities
* Spinal injuries
* Existing neurological conditions
* Pregnancy due to possible posture changes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Improvement in Cervical Range of Motion (ROM) | 6 Months
  Cervical Posture Improvement:
  Measured using craniovertebral angle (CVA) via digital photogrammetry to assess forward head posture correction.
  An increased CVA indicates an improvement in head and neck alignment.

SECONDARY OUTCOMES:
Neck Pain Intensity | 6months
  Evaluated using the Visual Analog Scale (VAS) for pain intensity before and after the intervention.
  A decrease in VAS score signifies reduced discomfort and muscle strain.

OTHER OUTCOMES:
Muscle Activation & Endurance | 6 months
  Assessed using the Deep Neck Flexor Endurance Test (DNFET) to measure the strength and endurance of deep cervical flexor muscles.
  Increased holding time in seconds reflects enhanced muscle activation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nadeem Ahmad, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Malakand, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No